CLINICAL TRIAL: NCT07179276
Title: Veno-arterial Carbon Dioxide Partial Pressure Difference (CO2gap) for Early Resuscitation of Septic Shock: A Multicenter Prospective Randomized Trial (CARBON)
Brief Title: Veno-arterial Carbon Dioxide Partial Pressure Difference (CO2gap) for Early Resuscitation of Septic Shock
Acronym: CARBON
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC N 2020 FUTIER
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Sepsis - to Reduce Mortality in the Intensive Care Unit; Septic Shock
Keywords: lactate; CO2 gap; resuscitation strategie; sepsis; hemodynamic therapy
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Masking Description: Data will be collected and entered into the electronic web-based case report form by trial or clinical trained personal blinded to the allocation group.
  Statistical analyses will be performed with the statistician blinded to the allocation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO2gap-guided resuscitation strategy (Experimental): CO2gap-guided resuscitation strategy aimed at maintaining central venous-to-arterial CO2 partial pressure difference (CO2gap) lower than 6 mmHg, using a sequential approach through a dedicated hemodynamic algorithm. Arterial and central venous blood samples will be drawn simultaneously and reassessed at 2 to 4-hour intervals
  Interventions: Procedure: CO2gap-guided resuscitation strategy
- Lactate level-guided resuscitation strategy (No Intervention): Lactate level-guided resuscitation strategy aimed at normalizing or decreasing lactate levels by 20% at 2 to 4-hour intervals, as per the surviving sepsis campaign guidelines.

INTERVENTIONS:
Procedure: CO2gap-guided resuscitation strategy — For patients assigned to the interventional arm, adherence to the algorithm will complement clinical practices in the following areas:
  * Blood sampling for venous blood gas analysis. Blood samples will be taken from an existing central venous catheter; central venous access is common clinical practice in critically ill patients.
  * The use of dobutamine and blood transfusions in patients showing signs of oxygen deficiency (both will be carried out in accordance with the intended use and conditions of current practice).
  Arms: CO2gap-guided resuscitation strategy

SUMMARY:
Sepsis is a dysregulated host response to infection that leads to life-threatening organ dysfunction and represents a major healthcare problem. Septic shock is the most severe form, characterized by increased capillary permeability and vasodilation, resulting in hypotension and tissue hypoxia. Early identification and treatment of tissue hypoperfusion are pivotal components of initial resuscitation to limit progression to multiple organ dysfunction and death. The 2021 Surviving Sepsis Guidelines recommend guiding initial resuscitation by targeting decreases in serum lactate levels in patients with elevated lactate. However, although elevated lactate levels may reflect tissue hypoxia, serum lactate is not a direct marker of tissue perfusion. Hyperlactatemia may be attributable to mechanisms other than tissue hypoperfusion, such as accelerated aerobic glycolysis driven by excessive β-adrenergic stimulation or impaired clearance (e.g., in liver failure).

The venous-to-arterial carbon dioxide partial pressure difference (CO₂ gap), which is inversely related to cardiac output, has been shown to reflect the adequacy of venous blood flow to remove CO₂ from tissues. The CO₂ gap is closely linked to microcirculatory blood flow during the early resuscitation phase of septic shock and may effectively identify persistent tissue hypoperfusion in shock states. A persistently high CO₂ gap during early resuscitation has been associated with significantly higher 28-day mortality and increased Sequential Organ Failure Assessment (SOFA) scores. Moreover, the CO₂ gap has been shown to respond to changes in cardiac output during inotrope infusion in patients with low blood flow, suggesting that its assessment could be useful for therapeutic adjustments. Therefore, there are compelling arguments to evaluate the usefulness of the CO₂ gap in guiding early resuscitation in patients with septic shock.

The investigators postulated that CO₂ gap-guided early resuscitation may be more effective in improving outcomes than lactate-guided resuscitation.

DETAILED DESCRIPTION:
Main objective: The aim of the CARBON trial is to compare a veno-arterial CO2 difference-guided resuscitation strategy (CO2gap-guided strategy) with a lactate level-guided resuscitation on mortality in adults intensive care unit (ICU) patients fulfilling the SEPSIS-3 criteria consensus definition.

HYPOTHESIS: The investigators hypothesized that a CO2gap-guided resuscitation strategy during early septic shock would reduce mortality compared with a lactate level-guided resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older AND
* Acutely admitted to a study ICU AND
* Primary diagnosis of septic shock according to the Sepsis-3 criteria and defined as:

  * A suspected or documented site of infection or positive blood culture AND
  * Acute increase of at least 2 points in the Sequential Organ Failure Assessment (SOFA) score consequent to the infection AND
  * Having a serum lactate level >2 mmol/l AND
  * Requirement of vasopressors (any dose of norepinephrine) to maintain mean arterial pressure (MAP) ≥65 mmHg despite adequate fluid resuscitation (at least 1L of IV fluid in the last 24 hours prior to screening)

Exclusion Criteria:

* Septic shock for more than 12 hours at the time of screening
* Primary cause of hypotension not due to sepsis (e.g., acute bleeding)
* Decision not to resuscitate (or to limit full care) or not to intubate taken before obtaining consent
* Death is deemed to be imminent or inevitable or patients with an underlying disease process with a life expectancy of less than 3 months
* Anticipated surgery during the first 24 hours after randomization
* Patient or their relatives' refusal to participate
* Patients participating in another RCT with interventions possibly compromising the primary outcome
* Prior enrollment in the CARBON trial
* Known to be pregnant.
* Legal protection (i.e., incompetence to provide consent and no guardian or incarceration)
* No affiliation with the French health care system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-12-09 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary end point is all-cause mortality at 28 days after randomization | Every day until Day 28

SECONDARY OUTCOMES:
Key secondary endpoints | Every day until Day 28
  Duration of septic shock (i.e., vasopressor use) up to Day 28
Key secondary endpoints | Every day until Day 90
  All-cause mortality at Day 90
Secondary Efficacy Endpoints | Every day until Day 28
  Vasopressor-free and inotrope-free days up to Day 28
Secondary Efficacy Endpoints | Every day until Day 28
  Renal replacement therapy-free days (excluding patients on renal replacement therapy at time of randomization) up to Day 28
Secondary Efficacy Endpoints | Every day until Day 28
  Mechanical ventilation-free days up to Day 28
Secondary Efficacy Endpoints | Every day until Day 28
  Duration of renal replacement therapy (excluding patients on renal replacement therapy at time of randomization) up to Day 28
Secondary Efficacy Endpoints | Every day until Day 28
  Duration of mechanical ventilation up to Day 28
Secondary Efficacy Endpoints | Every day until Day 7
  Incidence of new organ dysfunction (based on the SOFA score) up to Day 7
Secondary Efficacy Endpoints | Every day until Day 28
  ICU-free days up to Day 28
Secondary Efficacy Endpoints | Every day until Day 28
  ICU length of stay up to Day 28
Secondary Efficacy Endpoints | Every day until Day 28
  Hospital length of stay up to Day 28
Secondary Efficacy Endpoints | At Day 90 after randomization
  EuroQol 5 Dimensions, 5 Levels (EQ-5D-5L) :a measure of health-related quality of life at Day 90:
  The EQ-5D-5L score is analyzed using the utility value (global index score).
  In France, the score ranges from about -0.53 (health states considered worse than death) to 1.00 (full health).
  0.00 corresponds to a health state equivalent to death.
Secondary Safety Endpoints | Every day until Day 28
  Incidence of adverse events with specific emphasis on the incidence of ischemic (e.g., myocardial, stroke, intestinal, limb ischemia) and arrhythmia (excluding sinus tachycardia or sinus arrhythmia) events reported as having a reasonable possibility of a causal relationship with the study procedures

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Clermont-Ferrand Estaing, Clermont-Ferrand
  - CHU Clermont-Ferrand Gabriel Montpied, Clermont-Ferrand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le Gall JR, Lemeshow S, Saulnier F. A new Simplified Acute Physiology Score (SAPS II) based on a European/North American multicenter study. JAMA. 1993 Dec 22-29;270(24):2957-63. doi: 10.1001/jama.270.24.2957. PMID 8254858
- [Background] Levey AS, Becker C, Inker LA. Glomerular filtration rate and albuminuria for detection and staging of acute and chronic kidney disease in adults: a systematic review. JAMA. 2015 Feb 24;313(8):837-46. doi: 10.1001/jama.2015.0602. PMID 25710660
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Laterre PF, Berry SM, Blemings A, Carlsen JE, Francois B, Graves T, Jacobsen K, Lewis RJ, Opal SM, Perner A, Pickkers P, Russell JA, Windelov NA, Yealy DM, Asfar P, Bestle MH, Muller G, Bruel C, Brule N, Decruyenaere J, Dive AM, Dugernier T, Krell K, Lefrant JY, Megarbane B, Mercier E, Mira JP, Quenot JP, Rasmussen BS, Thorsen-Meyer HC, Vander Laenen M, Vang ML, Vignon P, Vinatier I, Wichmann S, Wittebole X, Kjolbye AL, Angus DC; SEPSIS-ACT Investigators. Effect of Selepressin vs Placebo on Ventilator- and Vasopressor-Free Days in Patients With Septic Shock: The SEPSIS-ACT Randomized Clinical Trial. JAMA. 2019 Oct 15;322(15):1476-1485. doi: 10.1001/jama.2019.14607. PMID 31577035
- [Background] STARRT-AKI Investigators; Canadian Critical Care Trials Group; Australian and New Zealand Intensive Care Society Clinical Trials Group; United Kingdom Critical Care Research Group; Canadian Nephrology Trials Network; Irish Critical Care Trials Group; Bagshaw SM, Wald R, Adhikari NKJ, Bellomo R, da Costa BR, Dreyfuss D, Du B, Gallagher MP, Gaudry S, Hoste EA, Lamontagne F, Joannidis M, Landoni G, Liu KD, McAuley DF, McGuinness SP, Neyra JA, Nichol AD, Ostermann M, Palevsky PM, Pettila V, Quenot JP, Qiu H, Rochwerg B, Schneider AG, Smith OM, Thome F, Thorpe KE, Vaara S, Weir M, Wang AY, Young P, Zarbock A. Timing of Initiation of Renal-Replacement Therapy in Acute Kidney Injury. N Engl J Med. 2020 Jul 16;383(3):240-251. doi: 10.1056/NEJMoa2000741. PMID 32668114
- [Background] Fergusson D, Aaron SD, Guyatt G, Hebert P. Post-randomisation exclusions: the intention to treat principle and excluding patients from analysis. BMJ. 2002 Sep 21;325(7365):652-4. doi: 10.1136/bmj.325.7365.652. No abstract available. PMID 12242181
- [Background] Hayes MA, Timmins AC, Yau EH, Palazzo M, Hinds CJ, Watson D. Elevation of systemic oxygen delivery in the treatment of critically ill patients. N Engl J Med. 1994 Jun 16;330(24):1717-22. doi: 10.1056/NEJM199406163302404. PMID 7993413
- [Background] Deis AS, Whiles BB, Brown AR, Satterwhite CL, Simpson SQ. Three-Hour Bundle Compliance and Outcomes in Patients With Undiagnosed Severe Sepsis. Chest. 2018 Jan;153(1):39-45. doi: 10.1016/j.chest.2017.09.031. Epub 2017 Oct 5. PMID 28987477
- [Background] Pruinelli L, Westra BL, Yadav P, Hoff A, Steinbach M, Kumar V, Delaney CW, Simon G. Delay Within the 3-Hour Surviving Sepsis Campaign Guideline on Mortality for Patients With Severe Sepsis and Septic Shock. Crit Care Med. 2018 Apr;46(4):500-505. doi: 10.1097/CCM.0000000000002949. PMID 29298189
- [Background] Seymour CW, Gesten F, Prescott HC, Friedrich ME, Iwashyna TJ, Phillips GS, Lemeshow S, Osborn T, Terry KM, Levy MM. Time to Treatment and Mortality during Mandated Emergency Care for Sepsis. N Engl J Med. 2017 Jun 8;376(23):2235-2244. doi: 10.1056/NEJMoa1703058. Epub 2017 May 21. PMID 28528569
- [Background] Creteur J, De Backer D, Vincent JL. A dobutamine test can disclose hepatosplanchnic hypoperfusion in septic patients. Am J Respir Crit Care Med. 1999 Sep;160(3):839-45. doi: 10.1164/ajrccm.160.3.9807029. PMID 10471606
- [Background] Teboul JL, Mercat A, Lenique F, Berton C, Richard C. Value of the venous-arterial PCO2 gradient to reflect the oxygen supply to demand in humans: effects of dobutamine. Crit Care Med. 1998 Jun;26(6):1007-10. doi: 10.1097/00003246-199806000-00017. PMID 9635647
- [Background] Mallat J, Pepy F, Lemyze M, Gasan G, Vangrunderbeeck N, Tronchon L, Vallet B, Thevenin D. Central venous-to-arterial carbon dioxide partial pressure difference in early resuscitation from septic shock: a prospective observational study. Eur J Anaesthesiol. 2014 Jul;31(7):371-80. doi: 10.1097/EJA.0000000000000064. PMID 24625464
- [Background] Vallee F, Vallet B, Mathe O, Parraguette J, Mari A, Silva S, Samii K, Fourcade O, Genestal M. Central venous-to-arterial carbon dioxide difference: an additional target for goal-directed therapy in septic shock? Intensive Care Med. 2008 Dec;34(12):2218-25. doi: 10.1007/s00134-008-1199-0. Epub 2008 Jul 8. PMID 18607565
- [Background] De Backer D. Detailing the cardiovascular profile in shock patients. Crit Care. 2017 Dec 28;21(Suppl 3):311. doi: 10.1186/s13054-017-1908-6. PMID 29297372
- [Background] Protti A, Masson S, Latini R, Fumagalli R, Romero M, Pessina C, Pasetti G, Tognoni G, Pesenti A, Gattinoni L, Caironi P. Persistence of Central Venous Oxygen Desaturation During Early Sepsis Is Associated With Higher Mortality: A Retrospective Analysis of the ALBIOS Trial. Chest. 2018 Dec;154(6):1291-1300. doi: 10.1016/j.chest.2018.04.043. Epub 2018 May 19. PMID 29787743
- [Background] Caironi P, Tognoni G, Masson S, Fumagalli R, Pesenti A, Romero M, Fanizza C, Caspani L, Faenza S, Grasselli G, Iapichino G, Antonelli M, Parrini V, Fiore G, Latini R, Gattinoni L; ALBIOS Study Investigators. Albumin replacement in patients with severe sepsis or septic shock. N Engl J Med. 2014 Apr 10;370(15):1412-21. doi: 10.1056/NEJMoa1305727. Epub 2014 Mar 18. PMID 24635772
- [Background] Mouncey PR, Osborn TM, Power GS, Harrison DA, Sadique MZ, Grieve RD, Jahan R, Harvey SE, Bell D, Bion JF, Coats TJ, Singer M, Young JD, Rowan KM; ProMISe Trial Investigators. Trial of early, goal-directed resuscitation for septic shock. N Engl J Med. 2015 Apr 2;372(14):1301-11. doi: 10.1056/NEJMoa1500896. Epub 2015 Mar 17. PMID 25776532
- [Background] ARISE Investigators; ANZICS Clinical Trials Group; Peake SL, Delaney A, Bailey M, Bellomo R, Cameron PA, Cooper DJ, Higgins AM, Holdgate A, Howe BD, Webb SA, Williams P. Goal-directed resuscitation for patients with early septic shock. N Engl J Med. 2014 Oct 16;371(16):1496-506. doi: 10.1056/NEJMoa1404380. Epub 2014 Oct 1. PMID 25272316
- [Background] ProCESS Investigators; Yealy DM, Kellum JA, Huang DT, Barnato AE, Weissfeld LA, Pike F, Terndrup T, Wang HE, Hou PC, LoVecchio F, Filbin MR, Shapiro NI, Angus DC. A randomized trial of protocol-based care for early septic shock. N Engl J Med. 2014 May 1;370(18):1683-93. doi: 10.1056/NEJMoa1401602. Epub 2014 Mar 18. PMID 24635773
- [Background] Neviere R, Chagnon JL, Teboul JL, Vallet B, Wattel F. Small intestine intramucosal PCO(2) and microvascular blood flow during hypoxic and ischemic hypoxia. Crit Care Med. 2002 Feb;30(2):379-84. doi: 10.1097/00003246-200202000-00019. PMID 11889315
- [Background] Vallet B, Teboul JL, Cain S, Curtis S. Venoarterial CO(2) difference during regional ischemic or hypoxic hypoxia. J Appl Physiol (1985). 2000 Oct;89(4):1317-21. doi: 10.1152/jappl.2000.89.4.1317. PMID 11007564
- [Background] Ronfle R, Lefebvre L, Duclos G, Rambaud R, Baumstarck K, Boucekine M, Daviet F, Baldesi O, Papazian L, Leone M. Venous-to-Arterial Carbon Dioxide Partial Pressure Difference: Predictor of Septic Patient Prognosis Depending on Central Venous Oxygen Saturation. Shock. 2020 Jun;53(6):710-716. doi: 10.1097/SHK.0000000000001442. PMID 31490355
- [Background] Bakker J, Vincent JL, Gris P, Leon M, Coffernils M, Kahn RJ. Veno-arterial carbon dioxide gradient in human septic shock. Chest. 1992 Feb;101(2):509-15. doi: 10.1378/chest.101.2.509. PMID 1735281
- [Background] Cuschieri J, Rivers EP, Donnino MW, Katilius M, Jacobsen G, Nguyen HB, Pamukov N, Horst HM. Central venous-arterial carbon dioxide difference as an indicator of cardiac index. Intensive Care Med. 2005 Jun;31(6):818-22. doi: 10.1007/s00134-005-2602-8. Epub 2005 Apr 1. PMID 15803301
- [Background] Vallet B, Pinsky MR, Cecconi M. Resuscitation of patients with septic shock: please "mind the gap"! Intensive Care Med. 2013 Sep;39(9):1653-5. doi: 10.1007/s00134-013-2998-5. Epub 2013 Jun 29. No abstract available. PMID 23812340
- [Background] Hernandez G, Ospina-Tascon GA, Damiani LP, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Granda-Luna V, Cavalcanti AB, Bakker J; The ANDROMEDA SHOCK Investigators and the Latin America Intensive Care Network (LIVEN); Hernandez G, Ospina-Tascon G, Petri Damiani L, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Cavalcanti AB, Bakker J, Hernandez G, Alegria L, Ferri G, Rodriguez N, Holger P, Soto N, Pozo M, Bakker J, Cook D, Vincent JL, Rhodes A, Kavanagh BP, Dellinger P, Rietdijk W, Carpio D, Pavez N, Henriquez E, Bravo S, Valenzuela ED, Vera M, Dreyse J, Oviedo V, Cid MA, Larroulet M, Petruska E, Sarabia C, Gallardo D, Sanchez JE, Gonzalez H, Arancibia JM, Munoz A, Ramirez G, Aravena F, Aquevedo A, Zambrano F, Bozinovic M, Valle F, Ramirez M, Rossel V, Munoz P, Ceballos C, Esveile C, Carmona C, Candia E, Mendoza D, Sanchez A, Ponce D, Ponce D, Lastra J, Nahuelpan B, Fasce F, Luengo C, Medel N, Cortes C, Campassi L, Rubatto P, Horna N, Furche M, Pendino JC, Bettini L, Lovesio C, Gonzalez MC, Rodruguez J, Canales H, Caminos F, Galletti C, Minoldo E, Aramburu MJ, Olmos D, Nin N, Tenzi J, Quiroga C, Lacuesta P, Gaudin A, Pais R, Silvestre A, Olivera G, Rieppi G, Berrutti D, Ochoa M, Cobos P, Vintimilla F, Ramirez V, Tobar M, Garcia F, Picoita F, Remache N, Granda V, Paredes F, Barzallo E, Garces P, Guerrero F, Salazar S, Torres G, Tana C, Calahorrano J, Solis F, Torres P, Herrera L, Ornes A, Perez V, Delgado G, Lopez A, Espinosa E, Moreira J, Salcedo B, Villacres I, Suing J, Lopez M, Gomez L, Toctaquiza G, Cadena Zapata M, Orazabal MA, Pardo Espejo R, Jimenez J, Calderon A, Paredes G, Barberan JL, Moya T, Atehortua H, Sabogal R, Ortiz G, Lara A, Sanchez F, Hernan Portilla A, Davila H, Mora JA, Calderon LE, Alvarez I, Escobar E, Bejarano A, Bustamante LA, Aldana JL. Effect of a Resuscitation Strategy Targeting Peripheral Perfusion Status vs Serum Lactate Levels on 28-Day Mortality Among Patients With Septic Shock: The ANDROMEDA-SHOCK Randomized Clinical Trial. JAMA. 2019 Feb 19;321(7):654-664. doi: 10.1001/jama.2019.0071. PMID 30772908
- [Background] Coopersmith CM, De Backer D, Deutschman CS, Ferrer R, Lat I, Machado FR, Martin GS, Martin-Loeches I, Nunnally ME, Antonelli M, Evans LE, Hellman J, Jog S, Kesecioglu J, Levy MM, Rhodes A. Surviving Sepsis Campaign: Research Priorities for Sepsis and Septic Shock. Crit Care Med. 2018 Aug;46(8):1334-1356. doi: 10.1097/CCM.0000000000003225. PMID 29957716
- [Background] Levy B. Lactate and shock state: the metabolic view. Curr Opin Crit Care. 2006 Aug;12(4):315-21. doi: 10.1097/01.ccx.0000235208.77450.15. PMID 16810041
- [Background] Casserly B, Phillips GS, Schorr C, Dellinger RP, Townsend SR, Osborn TM, Reinhart K, Selvakumar N, Levy MM. Lactate measurements in sepsis-induced tissue hypoperfusion: results from the Surviving Sepsis Campaign database. Crit Care Med. 2015 Mar;43(3):567-73. doi: 10.1097/CCM.0000000000000742. PMID 25479113
- [Background] Simpson SQ, Gaines M, Hussein Y, Badgett RG. Early goal-directed therapy for severe sepsis and septic shock: A living systematic review. J Crit Care. 2016 Dec;36:43-48. doi: 10.1016/j.jcrc.2016.06.017. Epub 2016 Jun 29. PMID 27546746
- [Background] Gu WJ, Zhang Z, Bakker J. Early lactate clearance-guided therapy in patients with sepsis: a meta-analysis with trial sequential analysis of randomized controlled trials. Intensive Care Med. 2015 Oct;41(10):1862-3. doi: 10.1007/s00134-015-3955-2. Epub 2015 Jul 8. No abstract available. PMID 26154408
- [Background] Yu B, Tian HY, Hu ZJ, Zhao C, Liu LX, Zhang Y, Zhu GJ, Wang LT, Wu XH, Li J. [Comparison of the effect of fluid resuscitation as guided either by lactate clearance rate or by central venous oxygen saturation in patients with sepsis]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2013 Oct;25(10):578-83. doi: 10.3760/cma.j.issn.2095-4352.2013.10.002. Chinese. PMID 24119693
- [Background] Tian HH, Han SS, Lv CJ, Wang T, Li Z, Hao D, Shang QM, Wang XZ. [The effect of early goal lactate clearance rate on the outcome of septic shock patients with severe pneumonia]. Zhongguo Wei Zhong Bing Ji Jiu Yi Xue. 2012 Jan;24(1):42-5. Chinese. PMID 22248751
- [Background] Lyu X, Xu Q, Cai G, Yan J, Yan M. [Efficacies of fluid resuscitation as guided by lactate clearance rate and central venous oxygen saturation in patients with septic shock]. Zhonghua Yi Xue Za Zhi. 2015 Feb 17;95(7):496-500. Chinese. PMID 25916923
- [Background] Jones AE, Shapiro NI, Trzeciak S, Arnold RC, Claremont HA, Kline JA; Emergency Medicine Shock Research Network (EMShockNet) Investigators. Lactate clearance vs central venous oxygen saturation as goals of early sepsis therapy: a randomized clinical trial. JAMA. 2010 Feb 24;303(8):739-46. doi: 10.1001/jama.2010.158. PMID 20179283
- [Background] Jansen TC, van Bommel J, Schoonderbeek FJ, Sleeswijk Visser SJ, van der Klooster JM, Lima AP, Willemsen SP, Bakker J; LACTATE study group. Early lactate-guided therapy in intensive care unit patients: a multicenter, open-label, randomized controlled trial. Am J Respir Crit Care Med. 2010 Sep 15;182(6):752-61. doi: 10.1164/rccm.200912-1918OC. Epub 2010 May 12. PMID 20463176
- [Background] Levy MM, Evans LE, Rhodes A. The Surviving Sepsis Campaign Bundle: 2018 update. Intensive Care Med. 2018 Jun;44(6):925-928. doi: 10.1007/s00134-018-5085-0. Epub 2018 Apr 19. No abstract available. PMID 29675566
- [Background] Vincent JL, De Backer D. Circulatory shock. N Engl J Med. 2013 Oct 31;369(18):1726-34. doi: 10.1056/NEJMra1208943. No abstract available. PMID 24171518
- [Background] Fleischmann C, Scherag A, Adhikari NK, Hartog CS, Tsaganos T, Schlattmann P, Angus DC, Reinhart K; International Forum of Acute Care Trialists. Assessment of Global Incidence and Mortality of Hospital-treated Sepsis. Current Estimates and Limitations. Am J Respir Crit Care Med. 2016 Feb 1;193(3):259-72. doi: 10.1164/rccm.201504-0781OC. PMID 26414292
- [Background] Liu V, Escobar GJ, Greene JD, Soule J, Whippy A, Angus DC, Iwashyna TJ. Hospital deaths in patients with sepsis from 2 independent cohorts. JAMA. 2014 Jul 2;312(1):90-2. doi: 10.1001/jama.2014.5804. No abstract available. PMID 24838355
- [Background] Seymour CW, Liu VX, Iwashyna TJ, Brunkhorst FM, Rea TD, Scherag A, Rubenfeld G, Kahn JM, Shankar-Hari M, Singer M, Deutschman CS, Escobar GJ, Angus DC. Assessment of Clinical Criteria for Sepsis: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):762-74. doi: 10.1001/jama.2016.0288. PMID 26903335
- [Background] Shankar-Hari M, Phillips GS, Levy ML, Seymour CW, Liu VX, Deutschman CS, Angus DC, Rubenfeld GD, Singer M; Sepsis Definitions Task Force. Developing a New Definition and Assessing New Clinical Criteria for Septic Shock: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):775-87. doi: 10.1001/jama.2016.0289. PMID 26903336
- [Background] Ospina-Tascon GA, Bautista-Rincon DF, Umana M, Tafur JD, Gutierrez A, Garcia AF, Bermudez W, Granados M, Arango-Davila C, Hernandez G. Persistently high venous-to-arterial carbon dioxide differences during early resuscitation are associated with poor outcomes in septic shock. Crit Care. 2013 Dec 13;17(6):R294. doi: 10.1186/cc13160. PMID 24330804
- [Background] Ospina-Tascon GA, Umana M, Bermudez WF, Bautista-Rincon DF, Valencia JD, Madrinan HJ, Hernandez G, Bruhn A, Arango-Davila C, De Backer D. Can venous-to-arterial carbon dioxide differences reflect microcirculatory alterations in patients with septic shock? Intensive Care Med. 2016 Feb;42(2):211-21. doi: 10.1007/s00134-015-4133-2. Epub 2015 Nov 17. PMID 26578172
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Angus DC, van der Poll T. Severe sepsis and septic shock. N Engl J Med. 2013 Aug 29;369(9):840-51. doi: 10.1056/NEJMra1208623. No abstract available. PMID 23984731
- See also: How Can We Use Tissue Carbon Dioxide Measurement as an Index of Perfusion? E. Futier, J.-L. Teboul, and B. Vallet — https://link.springer.com/chapter/10.1007/978-3-642-18081-1_33